CLINICAL TRIAL: NCT06723509
Title: Description of Patient Adherence to Heart Failure Remote Monitoring and Its Determinants
Acronym: TELE'IC
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-05Obs-CHRMT
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Remote Monitoring; Heart Failure Patients
Keywords: remote monitoring; heart failure patients; adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a monocentric cohort study, with retrospective data collection and prospective semi-structured interviews.

All patients who, since 2020, have received telemonitoring for heart failure after hospitalization at the CHR Metz-Thionville will be included. Patients will be informed of the study by e-mail, or by post if no e-mail is available. Data concerning their socio-demographic and clinical characteristics will be collected from the computerized patient record, and telerecording data will be extracted from the telerecording software.

Patients whose follow-up is still in progress will be monitored (=simple data collection) for 12 months, or until follow-up is terminated if necessary. Patients whose follow-up has been interrupted for less than a month at the start of the study (to avoid memory bias) or during the course of the study will be contacted by telephone by the IPA carrying out the telemonitoring, and offered, after oral consent, a semi-structured interview to investigate the reasons for the interruption.

DETAILED DESCRIPTION:
In 2022, the Caisse Primaire d'Assurance Maladie indicated that 'more than 1.5 million people suffer from heart failure, particularly the over-60s. Heart failure has a major impact on the quality of life of individuals and their families. It is the cause of 200,000 hospitalisations a year. With an ageing population, the incidence of heart failure is set to increase by 25% every four years over the next few years'.

In its WHITE PAPER, the Conseil National Professionnel Cardio Vasculaire recommended the day-to-day use of digital tools to monitor patients in the face of delays in consultations in towns and cities. According to the studies carried out, these 'delays (...) are such that they do not prevent 47.4% of patients from being admitted to hospital more than 15 days after the onset of the first symptoms. For a third of patients, this delay rises to more than 2 months'.

According to Brandon et al, in 2009 remote monitoring of patients with the implementation of call by an ABI reduces CI-related readmissions and this helps to improve patients' quality of life.However, they noted that this required 'further exploration of the role of the API in helping patients with CI achieve desired outcomes.'A 2022 study based on a multicentre randomised controlled trial showed that remote monitoring after hospitalisation improved survival in heart failure patients.

Other chronic pathologies are also monitored remotely, such as inflammatory arthritis.A prospective cohort study of 220 patients conducted by J. WIEGEL, published in 2022, looked at the profile of patients who did or did not adhere to remote monitoring of their condition.It was found that women discontinued this type of treatment more quickly. In conclusion, he wondered about the 'reasons why patients do not adhere to telemonitoring, as well as the reasons why they do'. He concluded by saying that these reasons 'must be studied in order to improve the adaptation of telemonitoring'.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Heart failure
* Having received telemonitoring for heart failure from the CHR
* Patient clearly informed about the research in progress
* Gave oral consent for telephone interview

Exclusion Criteria:

* Refusal to reuse data for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to break in remote monitoring (survival) | up to four years after start of remote monitoring
  Defined as the number of months of remote monitoring performed before interruption - no response from the patient after 6 weeks of reminders at a rate of 2 reminders per week, excluding justified absences. Cancellation of remote monitoring for any other reason will be considered a right censorship

SECONDARY OUTCOMES:
Proportion of patients who break off follow-up at 6 months | 6 months after start of remote monitoring
Proportion of patients who break off follow-up at 12 months | 12 months after start of remote monitoring
  Proportion of patients who break off follow-up
Proportion of patients who break off follow-up at 24 months | 24 months after start of remote monitoring
  Proportion of patients who break off follow-up
Break-off | up to four years after start of remote monitoring
  Mean time to break-off

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHR Metz Thionville Hopital de Mercy, Metz
  - CHR Metz-Thionville Hopital Bel Air, Thionville

IPD SHARING:
Plan to Share IPD: No